CLINICAL TRIAL: NCT04129684
Title: A Randomized Single-blind, Parallel-arm Multi-center Clinical Trial to Evaluate the Effectiveness and Safety of Lactobacillus Reuteri for Treatment of Periodontitis in a Chinese Population
Brief Title: A Clinical Trial to Evaluate the Effectiveness of Lactobacillus Reuteri for Periodontitis in a Chinese Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: West China College of Stomatology (Other); Peking University Third Hospital (Other); Hospital of Stomatology, Jilin University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-1015
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): SRP+BioGaia Prodentis oil drops and lozenges
  Interventions: Other: Probiotics
- Control group (Placebo Comparator): SRP+subgingival delivery of placebo and placebo lozenges
  Interventions: Other: Probiotics

INTERVENTIONS:
Other: Probiotics — subgingival delivery and lozenges

SUMMARY:
The aim of this study is to determine the efficacy of application of Lactobacillus Reuteri probiotics therapy on clinical improvement and on microbial shift in Chinese periodontitis patients.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease with a prevalence of 80% in Chinese adults, which is the main cause of tooth loss in adults. Periodontitis has also been demonstrated to be a risk factor for cardiovascular diseases, diabetes, and many other systemic diseases due to the host immune response elicited by periodontal pathogenic bacteria. In the last decade, probiotics therapy using Lactobacillus Reuteri has been applied for periodontitis patients in European countries. But no evidence has been provided for its effectiveness in a Chinese population. The aim of this study is to determine the efficacy of application of Lactobacillus Reuteri probiotics therapy on clinical improvement and on microbial shift in Chinese periodontitis patients. The influence of probiotics therapy on the host inflammatory cytokines levels in periodontitis patients with systemic diseases is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. Patients diagnosed with periodontitis clinically evident according to International Classification of Periodontal Diseases (2017) with periodontal probing depth ≥4mm, attachment loss of the most severe site in the adjacent area ≥3mm, and imaging bone loss more than 1/3 of the root length
3. Natural teeth remaining in the mouth≥ 14

Exclusion Criteria:

1. Patients with any other systemic diseases which likely to alter the progression and course of periodontitis, except coronary disease, diabetes or hypertension.
2. Patients with aggressive periodontitis.
3. Patients who received any periodontal treatment in the past 6 months
4. Pregnant or lactating women
5. Patients who smoke
6. Patients in the acute phase of an infectious disease
7. Patients taking bisphosphonate mediation
8. Patients who are on any probiotic, anticoagulants or antibiotic supplements for the past 3 months
9. Patients allergic to lactate products
10. Patients who are deemed uncooperative

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pocket Probing Depth(PPD) | at 3 months
  Distance from the base of the periodontal pocket to the gingival margin(mm)

SECONDARY OUTCOMES:
Change from baseline in Pocket Probing Depth | at baseline, 1, 6 months
  Distance from the base of the periodontal pocket to the gingival margin(mm)
Change from baseline in Clinical Attachment Level | at baseline, 1, 3 , 6 months
  Distance from the base of the periodontal pocket to the CEJ or other fixed reference point (mm)
Change from baseline in Rate of Bleeding on Probing | at baseline, 1, 3 , 6 months
  To evaluate the inflammation and bleeding of gingiva (%)
Number of microorganisms in periodontal pockets | at baseline, 1, 3 and 6 months
  To observe the effectiveness of the probiotic on periodontal microorganisms: P. gingivalis; A. actinomycetemcomitans; T. forsythia; T. denticola; P. intermedia; L. reuteri (CFU)
Contents of inflammatory cytokines in periodontal pockets and blood | at baseline, 1, 3 and 6 months
  To observe the effectiveness of the probiotic on systemic and local inflammation: TNF-α; IL-1β; IL-6; IL-8; IL-10；INF-γ (Pg/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Hangzhou, Zhejiang University, China

IPD SHARING:
Plan to Share IPD: Undecided